CLINICAL TRIAL: NCT02049944
Title: Increased Cefazolin (Ancef) Dosing for Prophylaxis During Cesarean Delivery in the Obese Population
Brief Title: Increased Cefazolin During Cesarean Delivery in Obese Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 186-13
Record Dates: First submitted 2014-01-24; First posted 2014-01-30 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Obesity, Morbid; Pregnancy; Infection; Cesarean Section
Keywords: Antibiotic Prophylaxis; Obesity; Obesity, Morbid; Pregnancy; Infection; Cesarean Section
MeSH Terms: conditions — Obesity; Obesity, Morbid; Infections | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefazolin (Experimental): All subjects undergoing elective term cesarean delivery will receive 3 grams of Cefazolin at least 30, but no more than 60 minutes prior to skin incision.
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Participants who are undergoing an elective cesarean section at term will receive 3 grams of Cefazolin at least 30, but no more than 60 minutes prior to skin incision administered through an intravenous line.
  Other Names: Ancef

SUMMARY:
The purpose of this study is to determine whether an increased prophylactic dose (3 grams) of cefazolin at the time of cesarean delivery has superior coverage in adipose tissue than the current established dosing of 2 grams. The tissue and serum concentration values, when using an increased prophylactic dose, can then be compared to our pilot study assays in hopes of determining an optimal dosing for the obese and morbidly obese populations undergoing cesarean delivery.

A previous study performed at University of California, Irvine (UCI) and Long Beach Memorial Medical Center/Miller Children's Hospital (LBMMC) showed that the standard dose of antibiotics (2 grams of cefazolin) did not provide adequate coverage for all organisms in the obese and extremely obese populations. The purpose of this research study is to evaluate whether in increased dose of antibiotics given before cesarean delivery (3 grams of cefazolin) will reach adequate levels in adipose (fat cells underneath the skin) and serum (blood) samples. In addition, researchers hope to evaluate if/how the mother's weight has an effect on the levels of antibiotics in the tissues (a group of similar cells).

This follow up study (prior study HS# 2009-7015 at UCI) will enroll obese (Body Mass Index (BMI) of 30-40) and morbidly obese (BMI >40) women to receive an increased dose of prophylactic cefazolin at time of scheduled cesarean delivery at both UCI and LBMMC. Researchers hope to enroll a total of 35 women overall.

DETAILED DESCRIPTION:
Study Design:

This is a follow-up to the original pilot study (HS# 2009-7015 at UCI/587-08 at LBMMC). This study is also designed to be a prospective, non-randomized, non-blinded trial of the effects of obesity on adequacy of antimicrobial (cefazolin) concentrations with increased doses (from 2 grams to 3 grams) of preoperative prophylactic antibiotics within adipose tissues at the time of cesarean delivery.

Inclusion Criteria:

• Patients at term (>37 weeks) undergoing a cesarean delivery at LBMMC and UCI.

Exclusion criteria:

* pre-gestational diabetes
* chronic hypertension
* collagen vascular disease
* renal impairment
* multiple gestation
* contraindications to cefazolin administration (known anaphylactic reaction to penicillin's or known cephalosporin allergy)
* any exposure to cephalosporins in one week prior to cesarean section
* need for emergent cesarean delivery or diagnosis of chorioamnionitis

Study Procedure:

All patients requiring cesarean delivery under non-emergent circumstances, as determined by their physician, will be approached for participation in study by co-investigators. They will be approached on Labor and Delivery during their intake evaluation on the day of their scheduled procedure. Based on published literature and preliminary power analysis we expect that each of the 2 study groups will need 1414 subjects to demonstrate statistically significant difference in antibiotic concentrations within adipose tissue. The two groups will consist of:

1. OBESE GROUP (BMI 30-40)
2. MORBIDLY OBESE GROUP (BMI >40)

   1. All subjects will receive cefazolin at least 30, but no more than 60 minutes prior to skin incision.
   2. At the time of cesarean delivery, the following tissue samples will be collected:

      * adipose tissue immediately following skin incision (prior to incision of the fascia) and
      * adipose tissue prior to skin closure
      * serum sample after skin incision but prior to completion of the operative procedure

Approximately 2 grams of tissue sampled from each site and 5 cc of blood will be required for analysis.

All samples will be collected by Dr. Swank, Dr. Wing or a physician who had previously been proctored in the proper tissue collecting techniques by either of the above mentioned investigators. Upon collection, tissue specimens will be blotted to remove residual blood and debris, weighed, and placed in a freezer (-80'C) until analysis. Serum samples will be drawn into red top tubes and immediately placed on wet ice. Immediately following completion of the surgery, they will then be centrifuged for 10 minutes at 3G (3200 rpm) and placed in a locked -80'C freezer until analysis.

Tissue and serum samples will then be sent to David P. Nicolau, PhD, FCCP, FIDSA, at the Center for Anti-Infective Research and Development, Hartford Hospital, Hartford, Connecticut. Samples will be batched and sent all together at the completion of study enrollment. Dr. Swank and the study nurse will be responsible for securely packing samples on dry ice and overnight shipping them to Dr. Nicolau. Once with Dr. Nicolau, the tissue samples will be homogenized and analyzed to determine zones of inhibition. The Cefazolin concentrations will be determined in the serum samples using a previously validated high-performance liquid chromatography method. 16 Tissues and serum will be sent without direct identifiers. Dr. Nicolau will not have access to the identity of the research subjects providing the samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients at term (>37 weeks) undergoing a cesarean delivery at Women's Pavilion at Miller Children's Hospital and University of California, Irvine.

Exclusion Criteria:

* pre-gestational diabetes
* chronic hypertension
* collagen vascular disease
* renal impairment
* multiple gestation
* contraindications to Cefazolin administration (known anaphylactic reaction to penicillin's or known cephalosporin allergy)
* any exposure to cephalosporins in one week prior to cesarean section
* need for emergent cesarean delivery or diagnosis of chorioamnionitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNulty, MD, Principal Investigator — MemorialCare Center for Women at Miller Children's Hospital Long Beach and Long Beach Memorial Medical Center; Deborah A Wing, MD, Principal Investigator — University of California, Irvine; Morgan Swank, MD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - MemorialCare Center for Women at Miller Children's Hospital Long Beach and Long Beach Memorial Medical Center, Long Beach, California
  - University of California, Irvine, Orange, California

RESULTS

PARTICIPANT FLOW:
Groups:
- 3g Cefazolin: Prospective cohort obese women receiving 3g prophylactic cefazolin 30-60 minutes prior to scheduled cesarean delivery
Period: Overall Study
Arm/Group | 3g Cefazolin
Started | 30
Obese (BMI 30-40kg/m^2) | 14
Extremely Obese (BMI >40kg/m^2) | 14
Completed | 28
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- 3g Cefazolin: 3g IV cefazolin given 30-60 minutes prior to skin incision
Arm/Group | 3g Cefazolin
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31.5 [26.5 to 36.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 18
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
preoperative hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 12.0 [11.4 to 12.6]
Average BMI [Mean (Standard Deviation); unit: kg/m2] — Population: these data were analyzed by BMI category, 14 obese and 14 extremely obese.
  kg/m2
    Obese, BMI 30-40kg/m^2: number analyzed (Participants) | 14
    Obese, BMI 30-40kg/m^2 | 33.82 (2.92)
    Extremely Obese, BMI >40kg/m^2: number analyzed (Participants) | 14
    Extremely Obese, BMI >40kg/m^2 | 45.03 (3.77)

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Minimal Inhibitory Concentrations Within Adipose and Serum Sampled at Time of Cesarean Delivery
Description: Primary Objective:
  To assess the effects of increased prophylactic doses of Cefazolin in the obese and morbidly obese populations undergoing cesarean delivery. Effects will be defined as the ability to reach the minimal inhibitory concentrations for gram-positive and gram-negative organisms in adipose tissue and serum at time of skin incision and skin closure as defined by the Clinical and Laboratory Standards Institute
Time Frame: Each participant is to be observed per routine operative and post-operative guidelines, inpatient for 3-4 days.
Population: participants were divided in BMI categories, 30-40kg/m2 and >40kg/m2.
Measure: Median (Inter-Quartile Range); unit: mg/g
Arm/Group | 3g Cefazolin
Number analyzed (Participants) | 28
mg/g
  BMI 30-40 3g: number analyzed (Participants) | 14
  BMI 30-40 3g | 22.4 [20.3 to 34.4]
  BMI >40 3g: number analyzed (Participants) | 14
  BMI >40 3g | 9.6 [7.6 to 15.8]
Statistical Analysis 1: Comparison: 3g Cefazolin; To detect the number of subjects who obtained a minimal inhibitory concentration (>4mg/ml) following increased 3g dose of cefazolin. Compare this number to the historical cohort who had received 2g of cefazolin (standard dosing); Test type: Other — we used t-test on the regression coefficient for the group indicator to test for differences in means categorical variables were evaluated using fisher's exact test of association linear regression for log transformed start adipose concentrations were calculated by dose specific group; Fisher Exact; Median Difference (Final Values) = 80

ADVERSE EVENTS:
Groups:
- 3g Cefazolin: 3g cefazolin provided via IV push 30-60 minutes prior to skin incision
Arm/Group | 3g Cefazolin
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No